CLINICAL TRIAL: NCT02162329
Title: Effects of Meditation on Cognitive Function and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0156; NCI-2015-00469 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2014-06-10; First posted 2014-06-12 (Estimated); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Cognitive function; Questionnaires; Surveys; Electroencephalography; EEG; Magnetic resonance imaging; fMRI; Tibetan meditation; Quality of life; QOL
MeSH Terms: conditions — Breast Neoplasms | interventions — Surveys and Questionnaires; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Healthy Control Group (Other): Healthy participants fill out several questionnaires asking questions about memory and concentration, mood, fatigue, how they have been feeling, and general quality of life. The questionnaires should take about 30 minutes to complete. Electroencephalography (EEG) and magnetic resonance imaging (fMRI) scan performed. These should take a total of about 90 minutes to complete.
  Interventions: Behavioral: Questionnaires; Procedure: Electroencephalography (EEG); Procedure: Magnetic Resonance Imaging (fMRI
- Tibetan Meditation Group (Experimental): Participants fill out several questionnaires at baseline, at completion of meditation classes, and at follow up visit. The forms should take about 30 minutes to complete. Participants complete computer tests to check memory and concentration taking about 20 minutes to complete. Electroencephalography (EEG) performed at baseline, at completion of classes, and at follow up visit. Participants have magnetic resonance imaging (fMRI) scan of brain at baseline, at completion of meditation classes, and at follow up visit. Tests, EEG, and fMRI should take a total of about 90 minutes to complete. Participants take part in up to 16 meditation classes for a total of 8 weeks. All sessions videotaped.
  Interventions: Behavioral: Questionnaires; Procedure: Electroencephalography (EEG); Procedure: Magnetic Resonance Imaging (fMRI; Behavioral: Meditation Classes
- Wait-List Group (Other): Participants fill out several questionnaires at baseline and at follow up visit. The forms should take about 30 minutes to complete. Participants complete computer tests to check memory and concentration taking about 20 minutes to complete. Tests, EEG, and fMRI should take a total of about 90 minutes to complete. Participants receive the standard of care for cancer patients.
  After 8 week follow up visit, Wait-List Group offered meditation program.
  Interventions: Behavioral: Questionnaires; Procedure: Electroencephalography (EEG); Procedure: Magnetic Resonance Imaging (fMRI

INTERVENTIONS:
Behavioral: Questionnaires — Participants fill out several questionnaires asking questions about memory and concentration, mood, fatigue, how they have been feeling, and general quality of life. The questionnaires should take about 30 minutes to complete.
  Meditation Group and Wait-List Group also complete questionnaires at follow up visit.
  Other Names: Surveys
Procedure: Electroencephalography (EEG) — Meditation Group and Wait-List Group: Electroencephalography (EEG) performed at baseline and at follow up visit. During EEG, 3 tests to check attention, short-term memory, and levels of emotions.
  Healthy Control Group: Electroencephalography (EEG) performed at study visit. During EEG, 3 tests to check attention, short-term memory, and levels of emotions.
  Other Names: EEG
Procedure: Magnetic Resonance Imaging (fMRI — Healthy Control Group: Magnetic resonance imaging (fMRI) scan performed.
  Meditation Group and Wait-List Group: Magnetic resonance imaging (fMRI) scan of brain performed at baseline and at follow up visit.
  Other Names: MRI
Behavioral: Meditation Classes — Participants take part in up to 16 meditation classes for a total of 8 weeks. All sessions videotaped.
  Arms: Tibetan Meditation Group

SUMMARY:
The goal of this research study is to test Tibetan meditation as a therapy to teach cancer patients to change their brain functioning and to improve quality of life. Researchers want to compare the cancer patients' outcomes to people who have never had cancer.

DETAILED DESCRIPTION:
Tibetan Meditation Program:

During the meditation program, you will learn several concepts such as focus, visualization, and sound. You will have up to 16 classes for 8 weeks. They should take about 60 minutes each.

First Study Visit:

If you choose to take part in this study, you will be asked to fill out several questionnaires. You will be asked questions about your memory and concentration, mood, fatigue, how you have been feeling, and your general quality of life. The forms should take about 30 minutes to complete.

You will complete some computer tests to check your memory and concentration. For example, you will be asked to remember a list of words and then be asked to recall them later. These tests should take about 20 minutes to complete.

You will then have an electroencephalography (EEG) done. An EEG checks a person's brainwaves. During the EEG, a snug cap which contains small electrodes will be placed on your head to measure the electrical patterns coming from the brain. This is like the way a doctor listens to your heart from the surface of your skin. During recording of the EEG, you will be asked to complete 3 tests to check your attention, short-term memory, and levels of emotions. For example, for one test you will use a use a keypad to choose a word's name that is a color (such as if the word "blue" written in the color red, the correct answer would be red).The EEG and tests will take about 45 minutes to one hour.

You will also have a functional magnetic resonance imaging (fMRI) scan of your brain. During the scan, you will lie down on your back with both arms extended by your sides. You will be fitted with earplugs and/or headphones to help dampen the noise caused by the scanner. The lights will also be dimmed. You will then lie still until the scan is over. The scan will take about 20 minutes.

The tests, EEG, and fMRI should take a total of about 90 minutes to complete.

Blood (about 1 tablespoon) will be drawn for tests to measure hormones and your immune system responses. This should take about 15 minutes.

All assessments will be performed at baseline and after the completion of classes.

Study Groups:

After the first study visit, you will be randomly assigned to 1 of 2 study groups. You will have about a 1 out of 2 chance of being assigned to each group. The groups are randomly assigned, but it is also based on other factors such as your age and the status of the disease.

Participants in the first group will take part in a meditation program. You will take part in up to 16 meditation classes for a total of 8 weeks. The meditation sessions may take place on any 2 days of the week at MD Anderson. During the meditation sessions, you will do deep breathing and visualization exercises and produce some sounds like "Ah." Each session will last about 60 minutes. A trained meditation instructor will teach the meditation sessions. Participants will be asked to continue daily meditation practice at home outside of the classes and will be given a CD to guide home practice. All sessions will be videotaped. This is so the researchers can keep track of the quality of the sessions. The audio and video files are digital and will be deleted after all the data are studied.

Participants in the second group will be in a wait-list group. You will continue to receive the standard of care for cancer patients, but you will not take part in the meditation program. You will be given the opportunity to take part in the meditation program and similar measures will be collected from you at similar times as that described below.

All participants must agree not to take part in any other meditation programs for as long as you take part in this study.

Follow-up Study Visit:

Within a week after the last meditation session (8 weeks after baseline), all participants will be asked to fill out a packet of questionnaires (like the ones at the first visit). It should take about 50 minutes to complete all of the questionnaires. You will have some tests to check your memory and concentration, similar to the tests you took at your initial visit. You will have another EEG and fMRI. You will have blood drawn.

After the 8 week follow-up, if you were in the meditation group your participation on this study will be over. If you were in the wait-list group you will be offered the meditation program and you will complete the same questionnaires as before. You will not have any more EEG or fMRI measurements or blood drawn.

You may receive reminder calls for each session and the follow-up study visit.

Length of Study:

If you are in the treatment group, you will be on study for up to 8 weeks. If you are in the waitlist group and decide to take meditation classes after the first 8 weeks, you may be on study for up to 16 weeks.

This is an investigational study.

Up to 140 participants will take part in this study. Up to 10 pilot participants without cancer will be take part in this study. Up to 40 participants without cancer and up to 80 patients will be enrolled. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Stage I - III female breast cancer patients who have undergone chemotherapy (either neoadjuvant or adjuvant) 6 - 60 months prior to recruitment
2. Report cognitive impairment since starting chemotherapy as assessed by four questions from the Functional Assessment of Cancer Therapy Cognitive Scale (FACT-Cog)
3. 35 to 65 years old
4. Able to read, write and speak English, Spanish, or Portuguese
5. Willing to come to MD Anderson Cancer Center (MDACC) or Hospital Israelita Albert Einstein (HIAE) for the meditation sessions and assessment sessions
6. Right handed (qEEG database comparison is specific to handedness. By requiring all participants be right handed, we will be consistent across EEG analysis.)
7. (PILOT PARTICIPANTS AND HEALTHY CONTROLS ONLY: Women with no history of cancer)
8. (PILOT PARTICIPANTS AND HEALTHY CONTROLS ONLY: No history of prior chemotherapy)
9. (PILOT PARTICIPANTS AND HEALTHY CONTROLS ONLY: 35 to 65 years old)
10. (PILOT PARTICIPANTS AND HEALTHY CONTROLS ONLY: Able to read, write, and speak English, Spanish, or Portuguese)
11. (PILOT PARTICIPANTS AND HEALTHY CONTROLS ONLY: Willing to come to MDACC and HIAE for the assessment session)
12. (PILOT PARTICIPANTS AND HEALTHY CONTROLS ONLY: Right handed)

Exclusion Criteria:

1. Diagnosis of a formal thought disorder (e.g., schizophrenia)
2. Any past neurologic insult that is known to affect brain function such as traumatic brain injury, dementia, encephalopathy, etc.
3. Mini-Mental State Examination score of 23 or below
4. Recurrent cancer
5. History of a neurological or psychological disorder that may interfere with the patient's ability to cooperate with study procedures
6. Factors contraindicated to fMRI
7. Any extreme mobility issues (e.g. unable to get in or out of a chair unassisted, extremity issues such as neuropathy that limits physical manipulation of objects
8. Regularly practiced meditation (greater than once per week) in the year prior to study enrollment
9. (PILOT PARTICIPANTS AND HEALTHY CONTROLS ONLY: Diagnosis of a formal thought disorder (e.g. schizophrenia))
10. (PILOT PARTICIPANTS AND HEALTHY CONTROLS ONLY: Mini-Mental State Examination score of 23 or below)
11. (PILOT PARTICIPANTS AND HEALTHY CONTROLS ONLY: Undergoing chemotherapy)
12. (PILOT PARTICIPANTS AND HEALTHY CONTROLS ONLY: Mini-Mental State Examination score of 23 or below)
13. (PILOT PARTICIPANTS AND HEALTHY CONTROLS ONLY: Any extreme mobility issues (e.g. unable to get in or out of a chair unassisted, extremity issues such as neuropathy that limits physical manipulation of objects)
14. (PILOT PARTICIPANTS AND HEALTHY CONTROLS ONLY: Primary caretaker of a cancer patient)
15. (PILOT PARTICIPANTS AND HEALTHY CONTROLS ONLY: Patients who have regularly practiced meditation (greater than once per week) in the year prior to study enrollment)

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2013-10-22 (Actual); Primary Completion 2022-10-18 (Actual); Study Completion 2022-10-18 (Actual)

PRIMARY OUTCOMES:
Changes in Cognitive Function | Assessed at baseline and 8 weeks after treatment
  Primary analyses based on difference scores of continuous variables measured at baseline and 8 weeks later. T tests or Wilcoxon two-sample tests used, depending on the distribution of the data. Reliable change index (RCI) used for the cognitive tasks. RCI based on standard error of measurement for each assessment and takes into account baseline levels of performance for any participant. A chi-square test used to compare the proportions of participants that fall into each classification in the meditation and control groups.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Cohen, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States
- Hospital Israelita Albert Einstein (HIAE), São Paulo, Brazil

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org